CLINICAL TRIAL: NCT01690117
Title: German Adaptation of Resources to Enhance Alzheimer's Caregiver Health
Brief Title: German Adaptation of REACH II
Acronym: GE-REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Hermann-Josef Gertz, Prof. Dr., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIA5-2512FSB552
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Dementia; Family Caregiver
Keywords: family caregiver; dementia; intervention; implementation
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GE-REACH-program (Experimental): GE-REACH-program
  Interventions: Behavioral: GE-REACH-program
- control group (No Intervention): usual care

INTERVENTIONS:
Behavioral: GE-REACH-program — The intervention program "Resources to Enhance Alzheimer's Caregivers Health -second step" (REACH II) is a multimodal, individualized and structured multi-component intervention program for family caregivers
  Arms: GE-REACH-program

SUMMARY:
The purpose of the present study is to adapt, to implement and to evaluate an support program for family caregivers of patients suffering from Alzheimers'Disease (AD). The intervention was comprehensive developed and successful evaluated in the USA and is called Resources to Enhance Alzheimers´Caregiver Health -second step (REACH II). To test the effectiveness of this German adaptation of REACH II the present implementation study is designed as randomized and controlled trial. Primary outcome is reducing family caregiver burden.

DETAILED DESCRIPTION:
Caring for elderly people with dementia imposes a heavy strain on care providers like family caregivers and puts them at risk of psychological and physical morbidity. A variety of psychosocial interventions have been developed which aim at improving caregiver emotional and physical health. These interventions differ in terms of treatment delivery (individual or group format) and content (education, symptom appraisal, problem solving, skill building, stress management or behavior modification). Systematic reviews and meta analyses have concluded that individualized programs have a greater impact than group interventions, and problem solving or behavior modification strategies are superior to education alone. Structured multi-component interventions may also reduce the risk of patients home admissions.

The intervention program "Resources to Enhance Alzheimer's Caregivers Health -second step" (REACH II) is a multimodal, individualized and structured multi-component intervention program for family caregivers and was successfully evaluated in a multisite, randomized and controlled trial in the USA. The overall objectives of REACH II are to identify and reduce modificable risk factors to enhance the well-being of the caregivers and to enhance the quality of care. It takes place at caregivers home and focuses on 5 domains that are important to caregivers: reducing depression, decreasing burden, improving self care, enhancing social support, and managing problem behaviours.

Since there is a lack of effective treatment programs for family caregivers of demented persons in the German Health system respectively care system the purpose of the present study is to adapt and to implement REACH II to the care system conditions of a medium-sized East German town (Leipzig). To test the effects of this adapted intervention program the present study is design as unisite, randomized and controlled trail. Primary outcome is reducing family caregiver burden.

ELIGIBILITY:
Inclusion criteria

* age 21 years or older
* living with or sharing cooking facilities with the care recipient
* providing care for a relative with a medical diagnosed Alzheimer disease or related disorder, vascular dementia or behavior variant frontotemporal dementia for at least 4 hours per day for at least the past 6 months

Exclusion criteria

* Involvment in another caregiver intervention
* actual psychiatric diagnosis of mental illness
* illness that would prevent 6 months of study participation
* forthcoming institutionalization of the person being cared.

Other requirements were logistic, including having a telephone, planning to remain in the geographic area for at least 6 months, and competency in German.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hermann-Josef Gertz, Prof. Dr., Principal Investigator — Klinik und Poliklinik für Psychiatrie der Universität Leipzig
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belle SH, Burgio L, Burns R, Coon D, Czaja SJ, Gallagher-Thompson D, Gitlin LN, Klinger J, Koepke KM, Lee CC, Martindale-Adams J, Nichols L, Schulz R, Stahl S, Stevens A, Winter L, Zhang S; Resources for Enhancing Alzheimer's Caregiver Health (REACH) II Investigators. Enhancing the quality of life of dementia caregivers from different ethnic or racial groups: a randomized, controlled trial. Ann Intern Med. 2006 Nov 21;145(10):727-38. doi: 10.7326/0003-4819-145-10-200611210-00005. PMID 17116917
- [Derived] Berwig M, Heinrich S, Spahlholz J, Hallensleben N, Brahler E, Gertz HJ. Individualized support for informal caregivers of people with dementia - effectiveness of the German adaptation of REACH II. BMC Geriatr. 2017 Dec 12;17(1):286. doi: 10.1186/s12877-017-0678-y. PMID 29233097
- [Derived] Heinrich S, Berwig M, Simon A, Janichen J, Hallensleben N, Nickel W, Hinz A, Brahler E, Gertz HJ. German adaptation of the Resources for Enhancing Alzheimer's Caregiver Health II: study protocol of a single-centred, randomised controlled trial. BMC Geriatr. 2014 Feb 12;14:21. doi: 10.1186/1471-2318-14-21. PMID 24520910

RESULTS

PARTICIPANT FLOW:
Groups:
- DeREACH-program: DeREACH-program
  DeREACH-program: The intervention program "Resources to Enhance Alzheimer's Caregivers Health -second step" (REACH II) is a multimodal, individualized and structured multi-component intervention program for family caregivers
- Control Group: usual care
  The informal caregivers of the control group only receive the standard supply of health care Services.
Period: Overall Study
Arm/Group | DeREACH-program | Control Group
Started | 47 | 45
Post-Measurement | 41 | 40
Completed | 31 | 31
Not Completed | 16 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DeREACH-program | Control Group | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (8.1) | 73.9 (8.2) | 73.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  Germany | 47 | 45 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Burden on the German Version of Zarit Caregiver Burden Interview (ZBI) (5-point Scale) at Month 6
Description: The ZBI is a validated , self-reported instrument assessing burden of caregivers of people with dementia over a undefined period of time. Possible scores range from 0 (no burden) to 88 (highest possible burden). Change = (month 6 - baseline score).
Time Frame: baseline and month 6
Population: The ZBI was compared between treatment groups using t-tests for independent samples on all randomised informal caregivers (intention-to-treat population). Several SPSS (Statistical Package for the Social Sciences ) - methods with missing value imputation were used, including expectation maximisation (EM) and multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DeREACH-program | Control Group
Number analyzed (Participants) | 41 | 40
units on a scale | -0.43 (8.41) | 7.05 (8.09)
Statistical Analysis 1: Comparison: DeREACH-program vs Control Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — The a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 7.47, 95% CI 2-sided [3.82 to 11.12], Standard Error of Mean 1.83

2. Primary Outcome: Change From Baseline in Burden on the German Version of Zarit Caregiver Burden Interview (ZBI) (5-point Scale) at Month 9
Description: The ZBI is a validated , self-reported instrument assessing burden of caregivers of people with dementia over a undefined period of time. Possible scores range from 0 (no burden) to 88 (highest possible burden). Change = (month 9 - baseline score).
Time Frame: baseline and month 9
Population: The ZBI was compared between treatment groups using t-tests for independent samples on all randomised informal caregivers (intention-to-treat population). Several SPSS methods with missing value imputation were used, including expectation maximisation (EM) and multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DeREACH-program | Control Group
Number analyzed (Participants) | 31 | 31
units on a scale | 2.67 (8.86) | 8.10 (8.58)
Statistical Analysis 1: Comparison: DeREACH-program vs Control Group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — The a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 5.43, 95% CI 2-sided [1.00 to 9.86], Standard Error of Mean 2.21

3. Secondary Outcome: Change From Baseline in Somatization on the Patient Health Questionaire - 15 Items (PHQ-15) - Module Somatization at Month 6
Description: PHQ-15 is a validated, self-reported instrument assessing somatization over the last 4-weeks time period. Possible scores range from 0 (no somatization) to 30 (most possible somatization). Change = (Month 6 Score - Baseline score)
Time Frame: baseline and 6 month
Population: The PHQ - 15 was compared between treatment groups using t-tests for independent samples on all randomised informal caregivers (intention-to-treat population). Several SPSS methods with missing value imputation were used, including expectation maximisation (EM) and multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DeREACH-program | Control Group
Number analyzed (Participants) | 41 | 40
units on a scale | -1.40 (3.48) | 1.59 (5.32)
Statistical Analysis 1: Comparison: DeREACH-program vs Control Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — The a priori threshold for statistical significance was 0.05. For the secondary outcomes inference statistics were explorative. Therefore the p-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 2.99, 95% CI 2-sided [1.01 to 4.97], Standard Error of Mean 1.00

4. Secondary Outcome: Change From Baseline in Somatization on the Patient Health Questionaire - 15 Items (PHQ-15) - Module Somatization at Month 9
Description: PHQ-15 is a validated, self-reported instrument assessing somatization over the last 4-weeks time period. Possible scores range from 0 (no somatization) to 30 (most possible somatization). Change = (Month 9 Score - Baseline score)
Time Frame: baseline and month 9
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DeREACH-program | Control Group
Number analyzed (Participants) | 31 | 31
units on a scale | -0.60 (4.00) | 1.10 (2.77)
Statistical Analysis 1: Comparison: DeREACH-program vs Control Group; Test type: Superiority or Other; p = 0.06, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 1.70, 95% CI 2-sided [-0.05 to 3.45], Standard Error of Mean 0.87

5. Secondary Outcome: Change From Baseline in Mental Health on the Patient Health Questionnaire - 4 Items (PHQ-4) (4-point Scale) at Month 6
Description: PHQ-4 is a validated, self-reported Instrument assessing mental health over a 2 - week period. Possible scores range from 0 (not ill) to 18 (worst possible mental illness). Change = (Month 6 Score - Baseline score)
Time Frame: baseline and month 6
Population: The PHQ-4 was compared between treatment groups using t-tests for independent samples on all randomised informal caregivers (intention-to-treat population). Several SPSS methods with missing value imputation were used, including expectation maximisation (EM) and multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group: DeREACH-program
  DeREACH-program: The intervention program "Resources to Enhance Alzheimer's Caregivers Health -second step" (REACH II) is a multimodal, individualized and structured multi-component intervention program for family caregivers
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 40
units on a scale | -0.66 (3.09) | 0.05 (3.05)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.30, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-0.65 to 2.07], Standard Error of Mean 1.22

6. Secondary Outcome: Change From Baseline in Mental Health on the Patient Health Questionnaire - 4 Items (PHQ-4) (4-point Scale) at Month 9
Description: PHQ-4 is a validated, self-reported Instrument assessing mental health over a 2 - week period. Possible scores range from 0 (not mental ill) to 18 (worst possible mental illness). Change = (Month 9 Score - Baseline score)
Time Frame: baseline and month 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 31
units on a scale | -0.29 (2.65) | 0.68 (3.67)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.24, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [-0.66 to 2.59], Standard Error of Mean 1.02

7. Secondary Outcome: Change From Baseline in Social Support on the ENRICHED-Social-Support-Instrument (ESSI) (5-point Scale) at Month 6
Description: ESSI is a validated, self-reported instrument assessing perceived social support of the caregivers over a undefined period of time. Possible scores range from 1 (no social support) to 25 (most possible social support). Change = (month 6 score - Baseline score)
Time Frame: baseline and month 6
Population: The ESSI was compared between treatment groups using t-tests for independent samples on all randomised informal caregivers (intention-to-treat population). Several SPSS methods with missing value imputation were used, including expectation maximisation (EM) and multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Group: The informal caregivers of the control group only receive the standard supply of health care Services.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 40
units on a scale | 0.66 (4.86) | 0.21 (4.45)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-2.50 to 1.62], Standard Error of Mean 1.04

8. Secondary Outcome: Change From Baseline in Social Support on the ENRICHED-Social-Support-Instrument (ESSI) (5-point Scale) at Month 9
Description: ESSI is a validated, self-reported instrument assessing perceived social support of the caregivers over a undefined period of time. Possible scores range from 1 (no social support) to 25 (most possible social support). Change = (month 9 score - Baseline score)
Time Frame: baseline and month 9
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 31
units on a scale | -0.55 (5.39) | -0.74 (4.12)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.88, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-2.63 to 2.25], Standard Error of Mean 8.86

9. Secondary Outcome: Change From Baseline in Psychological Quality of Life on the German Version of the Mental Component Summary of the General Health Questionaire Short Form 12 (SF-12) at Month 6
Description: SF-12 - mental component is a validated, self-reported instrument assessing psychological quality of live of the caregivers over the last four weeks time period. Possible scores range from 0 (lowest level of health) and 100 (highest level of health). Change = (Month 6 Score - Baseline score)
Time Frame: baseline and month 6
Population: The SF-12 -mental component was compared between treatment groups using t-tests for independent samples on all randomised informal caregivers (intention-to-treat population). Several SPSS methods with missing value imputation were used, including expectation maximisation (EM) and multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 40
units on a scale | 2.40 (8.70) | -2.53 (8.56)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Median Difference (Final Values) = -4.93, 95% CI 2-sided [-8.74 to -1.11], Standard Error of Mean 1.92

10. Secondary Outcome: Change From Baseline in Psychological Quality of Life on the German Version of the Mental Component Summary of the General Health Questionaire Short Form 12 (SF-12) at Month 9
Description: SF-12 is a validated, self-reported instrument assessing psychological and physical quality of live of the caregivers over the last four weeks time period. Possible scores range from 0 (lowest level of health) and 100 (highest level of health). Change = (Month 9 Score - Baseline score)
Time Frame: baseline and month 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 31
units on a scale | 3.87 (10.66) | -4.62 (8.16)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.49, 95% CI 2-sided [-13.31 to -3.66], Standard Error of Mean 2.41

11. Secondary Outcome: Change From Baseline in Physical Quality of Life on the German Version of the Physical Component Summary of the General Health Questionaire Short Form 12 (SF-12) at Month 6
Description: SF-12 is a validated, self-reported instrument assessing psychological and physical quality of live of the caregivers over the last four weeks time period. Possible scores range from 0 (lowest level of health) and 100 (highest level of health). Change = (Month 6 Score - Baseline score)
Time Frame: baseline and month 6
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 40
units on a scale | 2.60 (9.96) | -1.31 (7.71)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.05, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.91, 95% CI 2-sided [-7.86 to 0.04], Standard Error of Mean 1.98

12. Secondary Outcome: Change From Baseline in Physical Quality of Life on the German Version of the Physical Component Summary of the General Health Questionaire Short Form 12 (SF-12) at Month 9
Description: as for outcome 10
Time Frame: baseline and month 9
Population: The SF-12 - physical component was compared between treatment groups using t-tests for independent samples on all randomised informal caregivers (intention-to-treat population). Several SPSS methods with missing value imputation were used, including expectation maximisation (EM) and multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 31
units on a scale | -0.05 (9.59) | 0.19 (6.70)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.91, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-3.96 to 4.45], Standard Error of Mean 2.10

13. Secondary Outcome: Change From Baseline in Frequency of Problem Behavior on a German Version of the Frequency Subscale of the Revised Memory and Behavior Problem Checklist (RMBPC) - (5-point Scale) at Month 6
Description: RMBPC frequency subscale is a validated, proxy-reported instrument assessing the frequency of problem behavior of cognitively impaired persons over the last week time period. Possible scores range from 0 (never occured) and 96 (extremely often). Change = (Month 6 Score - Baseline score)
Time Frame: baseline and month 6
Population: The RMBPC - frequency subscale was compared between treatment groups using t-tests for independent samples on all randomised informal caregivers (intention-to-treat population). Several SPSS methods with missing value imputation were used, including expectation maximisation (EM) and multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 40
units on a scale | -1.62 (7.21) | 1.29 (5.89)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.05, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 2.90, 95% CI 2-sided [-0.01 to 5.81], Standard Error of Mean 1.47

14. Secondary Outcome: Change From Baseline in Frequency of Problem Behavior on a German Version of the Frequency Subscale of the Revised Memory and Behavior Problem Checklist (RMBPC) - (5-point Scale) at Month 9
Description: The frequency subscale of the RMBPC is a validated proxy-reported instrument assessing the frequency of problem behavior of cognitively impaired persons over the last week time period. Possible scores range from 0 (never occured) and 96 (extremely often). Change = (Month 9 Score - Baseline score)
Time Frame: baseline and month 9
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 31
units on a scale | 1.41 (8.02) | 3.09 (7.00)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 4.50, 95% CI 2-sided [0.68 to 8.33], Standard Error of Mean 1.91

15. Secondary Outcome: Change From Baseline in Strength of Reaction of Caregivers to Problem Behavior on a German Version of the Reaction Subscale of the Revised Memory and Behavior Problem Checklist (RMBPC) - (5-point Scale) at Month 6
Description: RMBPC reaction subscale is a validated self-reported instrument assessing the strength of reaction of caregivers to problem behavior of cognitively impaired persons over the last week time period. Possible scores range from 0 (no reaction) and 96 (extremely strong reaction). Change = (Month 6 Score - Baseline score)
Time Frame: baseline and month 6
Population: The RMBPC reaction subscale was compared between treatment groups using t-tests for independent samples on all randomised informal caregivers (intention-to-treat population). Several SPSS methods with missing value imputation were used, including expectation maximisation (EM) and multiple imputations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 41 | 40
units on a scale | -5.46 (7.26) | 2.34 (6.38)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -4.53, 95% CI 2-sided [-8.40 to -0.65], Standard Error of Mean 1.95

16. Secondary Outcome: Change From Baseline in Strength of Reaction of Caregivers to Problem Behavior on a German Version of the Reaction Subscale of the Revised Memory and Behavior Problem Checklist (RMBPC) - (5-point Scale) at Month 9
Description: RMBPC reaction subscale is a validated self-reported instrument assessing the strength of reaction of caregivers to problem behavior of cognitively impaired persons over the last week time period. Possible scores range from 0 (no reaction) and 96 (extremely strong reaction). Change = (Month 9 Score - Baseline score)
Time Frame: baseline and month 9
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 31 | 31
units on a scale | -6.17 (7.87) | 3.24 (7.00)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 7.80, 95% CI 2-sided [4.78 to 10.83], Standard Error of Mean 1.52

ADVERSE EVENTS:
Groups:
- Intervention Group; Control Group: Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No